CLINICAL TRIAL: NCT01445405
Title: Phase I Study of Bortezomib and Cetuximab Without or With Cisplatin in Combination With Radiation Therapy for Advanced Head and Neck Cancer
Brief Title: Radiation Therapy and Bortezomib and Cetuximab With or Without Cisplatin to Treat Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080071; 08-C-0071
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-02-08

CONDITIONS: Carcinoma, Squamous; Head and Neck Cancer; Oral Cancer; Laryngeal Cancer; Pharyngeal Cancer
Keywords: Proteasome; Bortezomib; NF-kappaB; Cetuximab; Epidermal Growth Factor; Head and Neck Cancer; Squamous Cell Carcinoma; Oral Cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms; Mouth Neoplasms; Laryngeal Neoplasms; Pharyngeal Neoplasms | interventions — Bortezomib; Cetuximab; Cisplatin; Radiotherapy

INTERVENTIONS:
Drug: Bortezomib (Velcade, PS-341)
Drug: Cetuximab
Drug: Cisplatin
Procedure: Radiation Therapy

SUMMARY:
Background:

Bortezomib acts on molecules in head and neck cancer cells that are important for the cells growth and survival. The drug may help make the cancer more sensitive to radiation and other chemotherapy drugs.

Cetuximab is a monoclonal antibody that has increased the effectiveness of radiation treatment in patients with head and neck cancer in clinical trials.

Cisplatin has shrunk head and neck cancers and improved treatment response and survival when combined with radiation treatment.

Objectives:

To determine the highest safe dose of bortezomib when combined with cetuximab without or with cisplatin and with radiation in patients with advanced head and neck cancer.

To examine the benefits and side effects of these drug combinations with radiation in patients with advanced head and neck cancer.

Eligibility:

Patients 18 years of age and older with advanced Stage IV head and neck cancer who have not previously had neck radiation.

Design:

Patients will be assigned sequentially to one of two treatment groups: Group A receives bortezomib and cetuximab beginning the week before, and for the duration of, radiation therapy; Group B receives bortezomib, cetuximab and cisplatin beginning the week before, and for the duration of, radiation therapy.

* Cetuximab is given as a 2-hour infusion through a vein (intravenously, IV) for the first dose and then over 1 hour for subsequent weekly doses.
* Bortezomib is given as an injection into a vein over about 5 seconds, twice a week for 2 weeks, followed by a 1-week rest for a total of three 3-week treatment cycles during radiation.
* Cisplatin is given in once a week as a 1-hour IV infusion
* Radiation therapy is given 5 days a week for 7 to 8 weeks.

Post-treatment follow-up:

* Until 2 weeks after treatment ends, patients are followed once a week including a physical examination, review of treatment side effects, and blood tests.
* For 2 months after treatment ends, patients may need to return to the hospital for medical evaluation and supportive care, depending on their condition.
* 8-weeks after treatment ends, patients return for evaluation with a history and physical examination; blood tests; ear, nose and throat evaluation and endoscopy; CT or MRI scan, or both, of the neck and chest; and, if indicated, a PET scan....

DETAILED DESCRIPTION:
Background:

* Advanced squamous cell carcinoma involving the head and neck (SCCHN) has a mortality exceeding 50 percent and significant impact on function and quality of life.
* Treatment of locally advanced SCCHN with anti-Epidermal Growth Factor Receptor (EGFR) antibody cetuximab (Erbitux or C225) or DNA damaging agent cisplatin concurrent with radiation therapy (RT) have shown improvements in response, survival, and organ preservation, of approximately10-20 percent over RT alone. The combination of cetuximab, cisplatin and RT is currently under investigation as the next standard for concurrent chemo-RT for patients with SCCHN.
* Cetuximab inhibits EGFR, which is overexpressed by approximately 90 percent of SCCHN and is associated with decreased patient survival. EGFR contributes to activation of the Mitogen Activated Protein Kinase (MAPK) and Signal Transduction and Activating Transcription Factor (STAT3) pathways, which promote induction of genes involved in cell proliferation and survival.
* Recently, the Nuclear Factor-kappaB (NF-kB) pathway has been shown to be an independent pathway important for altered expression of prosurvival genes, the malignant phenotype, and prognosis.
* Proteasome inhibitor bortezomib (Velcade, PS-341) can inhibit NF-kB and target genes, as well as increase expression of tumor suppressor genes such as p53 in SCCHN. Bortezomib in combination with RT, cetuximab or cisplatin induces greater cytotoxic effects in cancer cells than these treatments individually in preclinical studies.
* In this phase I trial we will determine the feasibility of administering bortezomib concurrently with cetuximab and RT, and cetuximab, cisplatin and RT. We hypothesize that bortezomib can be given with these combinations with an acceptable toxicity profile and a maximum tolerated dose (MTD) that demonstrates clinical activity and effects on NF-kB, MAPK and STAT3 pathway signaling and apoptosis in SCCHN.

Specific Objectives:

Primary Objectives

-To evaluate the feasibility and toxicities of combining the proteasome inhibitor bortezomib with cetuximab, or cetuximab and cisplatin concurrent with radiation for therapy of patients with advanced squamous cell carcinoma of the head and neck (SCCHN), and to identify the MTD for bortezomib for further clinical phase 2 development.

Secondary Objectives

-To evaluate the objective response rate, progression-free survival and overall survival with the above regimen.

To determine the effects of bortezomib with cetuximab, or bortezomib, cetuximab with cisplatin to inhibit activation of the NF-kB, EGFR, MAPK, and STAT3 signal pathways, expression of pro-survival and pro-angiogenesis genes regulated by these pathways, and effects on proliferation, apoptosis and angiogenesis.

Eligibility:

-Patients with advanced Stage IV SCCHN, without history prior neck radiation, for whom concurrent chemo-RT is an option.

Design:

* All patients will receive standard RT to a total dose of 70 Gy, in 2 Gy/day fractions, 5 days/week, concurrent with either bortezomib and cetuximab, or bortezomib, cetuximab and cisplatin.
* Bortezomib will be given following a dose escalation schema (3 dose levels of 0.7, 1 and 1.3 mg/m2/dose) IV twice weekly for the first two weeks of three 21-day cycles which each include a 1 week break, starting the week prior to RT initiation and for a total of 7-8 weeks.
* In group A, patients with receive bortezomib, cetuximab and RT, and in group B, bortezomib, cetuximab, cisplatin and RT.
* Previously established MTDs will be used for weekly administration of cetuximab (400mg/m2 initially and then 250 mg/m(2) IV weekly), and cisplatin (30mg/m(2) IV weekly).
* Cetuximab or cetuximab and cisplatin will be given with the first dose of bortezomib the week prior to RT and continue weekly during RT (7-8 weekly doses). Drug therapy will not be given after RT completion.
* Groups A will accrue before group B, to identify the MTD for the combination of bortezomib, cetuximab and RT, and then bortezomib, cetuximab, cisplatin and RT, for expansion and phase 2 development.
* Serum and blood will be collected for study of potential proteomic and genetic markers of drug sensitivity and effects, and tumor response and recurrence, within 2 weeks pretreatment and days 5, 12 of bortezomib cycle 1, and day 12 of cycles 2 and 3. Serum will be collected thereafter every 3 months up to 24 months.
* Optional tumor and/or skin biopsies will be performed within 2 weeks before start of treatment and on day 5 of the first week during treatment with drugs alone, and on day 12 after start of RT for correlative studies of the combined effects of bortezomib with cetuximab, or bortezomib cetuximab and cisplatin on signal pathway activation, apoptosis and other markers, without and with RT. (Details of correlative studies). Patients will be evaluated by CT and FDG-PET pre-treatment and for response 8 weeks post-RT using WHO RECIST criteria.
* The study design and sample size is Phase 1, 3-6 patients per dose level to establish the MTD. An additional 6-10 patients (in each group) will be treated at the MTD in order further assess toxicity, response and molecular correlatives. The anticipated sample size is between 6 and 46.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Histologically or cytologically confirmed squamous cell carcinoma, including variants, or undifferentiated/poorly differentiated carcinoma of the head and neck (any site, except nasopharynx).
2. Previously untreated stage IV disease (AJCC staging system, 6th edition), or,
3. Patients with residual disease or regional recurrence of head and neck cancer after surgery and/or chemotherapy, but with no prior bortezomib, EGFR inhibitor therapy or head and neck radiotherapy. All such patients should be eligible to receive full dose radiation therapy, and must be evaluated and accepted for treatment by a Radiation Oncologist. Prior cisplatin is allowed if administered greater than 3 months earlier.
4. Patients with no clinically measurable distant disease, or those with asymptomatic small distant lesions outside the radiation field of less than or equal to 3cm individual or aggregate diameter, but for whom palliation of local and regional disease is clinically warranted will be eligible.
5. Any number of other prior systemic therapies is allowed. Patients must have fully recovered from the effects of any prior surgery, or chemotherapy. A minimum time period of 4 weeks (6 weeks for nitrosoureas or mitomycin C) should elapse between the completion of prior chemotherapy and enrollment in the study.
6. Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of bortezomib in combination with cetuximab or cisplatin and radiation in patients <18 years of age, and head and neck cancer in children is exceedingly rare, except for those with disorders of DNA damage repair, bone marrow or transplant immunosuppression likely to have lower tolerance to these drugs and RT, children are excluded from this study.
7. ECOG performance status 0-1 (Karnofsky greater than or equal to 70 percent).
8. Patients must have normal organ and marrow function as defined below:

   * absolute neutrophil count greater than or equal to 1,500/mcL
   * platelets greater than or equal to 100,000/mcL
   * total bilirubin within normal institutional limits, except for patients with Gilberts syndrome, with increased indirect bilirubin less than or equal to 3 mg/dL
   * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 times institutional upper limit of normal
   * creatinine within normal institutional limits

   OR

   -creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.
9. The effects of bortezomib on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must have agreed to use adequate contraception (hormonal or barrier method of birth control; prior vasectomy; tubal ligation or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
10. Adequate cognitive and neurologic function to protect against and detect and report toxicities experienced, and to understand and to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Patients with previously untreated nasopharyngeal cancer (any stage) will be excluded, but patients with recurrent nasopharyngeal carcinoma will be eligible.
2. Prior treatment with radiation to the head and neck, or systemic EGFR inhibitors or bortezomib is not allowed.
3. Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
4. Patients may not be receiving any other investigational agents.
5. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to bortezomib, cetuximab, cisplatin or other agents used in study.
7. Patients with greater than or equal to grade 2 peripheral sensory neuropathy because bortezomib can cause irreversible worsening and a painful type of chemotherapy associated peripheral neuropathy.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Pregnant women are excluded from this study because bortezomib, cetuximab and cisplatin have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with bortezomib, cetuximab and cisplatin, breastfeeding should be discontinued if the mother is treated with bortezomib, cetuximab and cisplatin. These potential risks may also apply to other agents used in this study.
10. HIV-positive patients or patients on any antiretroviral therapy are ineligible because of the potential for possible pharmacodynamic interactions with bortezomib, cetuximab and cisplatin, particularly bone marrow and mucosal toxicity, which could affect the MTD. These patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-02-05; Primary Completion 2010-08-27 (Actual); Study Completion 2010-08-27 (Actual)

PRIMARY OUTCOMES:
Evaluate feasibility/toxicities of combining proteasome inhibitor bortezomib with cetuximab without/with cisplatin concurrent with radiation for therapy of Pts with advanced SCCHN, and identify MTD for bortezomib for further clinical phase 2 dev...

SECONDARY OUTCOMES:
1) Evaluate objective response rate, progression-free survival/overall survival with the above regimen. 2) Determine effects of bortezomib with cetuximab or with cetuximab/ cisplatin to inhibit activation of NF-kB, EGFR, MAPK, and STAT3 signal p...

CONTACTS AND LOCATIONS:
Overall Officials: Carter Van Waes, M.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Kotwall C, Sako K, Razack MS, Rao U, Bakamjian V, Shedd DP. Metastatic patterns in squamous cell cancer of the head and neck. Am J Surg. 1987 Oct;154(4):439-42. doi: 10.1016/0002-9610(89)90020-2. PMID 3661849
- [Background] Hong WK, Lippman SM, Itri LM, Karp DD, Lee JS, Byers RM, Schantz SP, Kramer AM, Lotan R, Peters LJ, et al. Prevention of second primary tumors with isotretinoin in squamous-cell carcinoma of the head and neck. N Engl J Med. 1990 Sep 20;323(12):795-801. doi: 10.1056/NEJM199009203231205. PMID 2202902